CLINICAL TRIAL: NCT04123353
Title: Reproducibility of Brain Volume and Lesion Measurements in Multiple Sclerosis: a Scan-Rescan Sub-Study of Multiple Sclerosis Partners Advancing Technology and Health Solutions (MS PATHS)
Brief Title: Scan-Rescan Sub-Study of MS PATHS
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 888MS004
Record Dates: First submitted 2019-09-24; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this sub-study is to calculate the reproducibility and other technical performance measures of various magnetic resonance imaging (MRI) image analysis algorithms in order to assess their suitability for detecting changes due to multiple sclerosis (MS) in a real-world setting in participants with MS. The secondary objective of this sub-study is to use the primary endpoint results to calibrate measurements across scanners within each MS PATHS center.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants (or participant's legal representative) has the ability to understand the purpose and risks of the sub-study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and l local participant privacy regulations.
* Diagnosis of relapse-onset MS (relapsing-remitting or secondary progressive).
* First MS symptom within the past 1 to 30 years.

Key Exclusion Criteria:

* Initiation of any MS disease-modifying treatment within 4 weeks prior to Visit 1.
* Steroid treatment or suspected MS relapse within 6 weeks prior to Visit 1.

Note: Other protocol specified inclusion and exclusion criteria may apply.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potential participants will be participants with MS enrolled in Study 888MS001 who have varying levels of disease severity and symptom duration.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-02-11 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Overall Reproducibility of Brain Volume | Baseline up to Day 7
Overall Reproducibility of Lesions | Baseline up to Day 7
Intrascanner Reproducibility of Brain Volume | Baseline up to Day 7
Intrascanner Reproducibility of Lesions | Baseline up to Day 7
Interscanner Reproducibility of Brain Volume | Baseline up to Day 7
Interscanner Reproducibility of Lesions | Baseline up to Day 7
Intra-class Correlation Coefficients (ICCs) Across Repeated Magnetic Resonance Imaging (MRI) for Brain Lesions | Baseline up to Day 7
Kappa Coefficients Across Expert Manual Segmentation for Brain Lesions | Baseline up to Day 7
Sensitivity and Specificity for Lesion Detection | Baseline up to Day 7

SECONDARY OUTCOMES:
Correlation Coefficients of Equation Parameters for Models to Map Brain Volume and Lesion Measurements between Scanners | Baseline up to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (3):
- United States (3):
  - Research Site, Baltimore, Maryland
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio